CLINICAL TRIAL: NCT05645679
Title: Efficacy and Safety of HYbrid Argon Plasma Coagulation Technique in Patients With Barrett's Esophagus-Related Dysplasia: a Multicenter Italian Prospective stuDy
Brief Title: Efficacy and Safety of HYbrid Argon Plasma Coagulation Technique in Patients With Barrett's Esophagus-Related Dysplasia
Acronym: HYBRID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2858
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-01

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Hybrid Argon Plasma Coagulation System — Hybrid Argon Plasma Coagulation System

SUMMARY:
Background Barrett's esophagus (BE) is defined by AGA as "a change in the esophageal epithelium of any length that can be recognized at upper endoscopy and is confirmed to have intestinal metaplasia by biopsy". It is a pre-malignant condition and may progress to low grade dysplasia, high grade dysplasia and ultimately esophageal adenocarcinoma which has poor prognosis with a 5-year survival rate of only 5-20%.Radiofrequency ablation (RFA) is a standard modality and well-studied endoscopic treatment for dysplastic BE. While the rate of complete eradication of dysplasia has been reported to be between 78% - 94% with RFA, the rate of complications associated with this procedure has been reported to be as high as 19.1%, and the costs are high. In a randomized clinical trial in patients with BE and low-grade dysplasia by Phoa et al in 2014, 68 patients underwent radiofrequency ablation therapy with a median of three ablation sessions per patient while 68 patients were randomized to endoscopic surveillance. In this study, a total of 13 patients (19.1%) experienced an adverse event in the treatment group versus no adverse events in the control group. Eight patients (11.8%) developed esophageal strictures which required a median of one dilation, three patients were noted to have small mucosal lacerations, one patient developed retrosternal pain treated with analgesics while one patient developed abdominal pain requiring hospitalization and treatment with analgesia. Several other studies have reported the rate of complications ranging between 5% to 19.1% and stricture formation being the most common among them. Hybrid argon plasma coagulation (H-APC) is a newer technique that involves submucosal fluid injection prior to performing APC. The injection of solutions (e.g., 0.9% sodium chloride solution (normal sterile saline) with or without supplementation of epinephrine, methylcellulose solution, hydroxyethyl starch, hyaluronic acid, autologous blood or blood substitute fluids) into the submucosa to limit the depth of thermal injury has been established both in pre-clinical studies for different tissues of the gastrointestinal tract and in the clinical practice for EMR and ESD, respectively.

ELIGIBILITY:
Inclusion Criteria:

- Patients with histopathologically confirmed LGD or HGD, or residual BE (Prague Classification ≤C3 / ≤M5) after endoscopic resection of a focal lesion containing LGD, HGD or early (≤T1sm1) cancer in the participating centres are eligible for study participation.

Exclusion Criteria:

* Younger than 18 years of age at time of consent
* Esophageal stenosis preventing advancement of a therapeutic endoscope
* Prior distal oesophagectomy
* Previous ablation therapy of the esophagus
* Active oesophagitis grade B or higher (patients can be included after appropriate treatment of reflux oesophagitis)
* History of oesophageal varices
* Achalasia
* Severe medical comorbidities precluding endoscopy
* Uncontrolled coagulopathy
* Pregnant or planning to become pregnant during period of study participation
* Life expectancy ≤2 years, as judged by the site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histopathologically confirmed LGD or HGD, or residual BE (Prague Classification ≤C3 / ≤M5) after endoscopic resection of a focal lesion containing LGD, HGD or early (≤T1sm1) cancer in the participating centres are eligible for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Hybrid Argon Plasma Coagulation Technique | 2 years
  percentage of patients with complete eradication of all Barrett's epithelium on endoscopy and CE-IM in all biopsies obtained at the first follow-up endoscopy after the maximum of 5 treatment sessions (and escape treatment(s) if necessary).
  the percentage of patients with CE-D in all biopsies obtained at the first follow-up endoscopy after the maximum of 5 treatment sessions (and escape treatment(s) if necessary).

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Massimi D, Maselli R, Pecere S, Spada C, Andrisani G, Di Matteo FM, La Terra A, Coppola F, Capogreco A, De Sire R, Alfarone L, Menini M, Spadaccini M, Hassan C, Repici A. Efficacy and safety of H-APC in Barrett's esophagus: Italian prospective multicenter study. Endosc Int Open. 2025 Feb 26;13:a25318227. doi: 10.1055/a-2531-8227. eCollection 2025. PMID 40018075